CLINICAL TRIAL: NCT01903993
Title: A Phase II, Open-label, Multicenter, Randomized Study to Investigate the Efficacy and Safety of MPDL3280A (Anti-PD-L1 Antibody) Compared With Docetaxel in Patients With Non-Small Cell Lung Cancer After Platinum Failure
Brief Title: A Randomized Phase 2 Study of Atezolizumab (an Engineered Anti-PDL1 Antibody) Compared With Docetaxel in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Failed Platinum Therapy - "POPLAR"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28753; 2013-001142-34 (EudraCT Number)
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; atezolizumab

ARMS (2):
- Docetaxel (Active Comparator): Participants received docetaxel 75 milligram per meter square (mg/m^2) administered intravenously on Day 1 of each 21 day cycle until disease progression or unacceptable toxicity or death.
  Interventions: Drug: Docetaxel
- Atezolizumab (Experimental): Participants were administered atezolizumab intravenously on Day 1 of each 21 day cycle at a fixed dose of 1200 mg. Atezolizumab treatment were to continued as long as participants were experiencing clinical benefit as assessed by the investigator.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Docetaxel — Participants received starting dose of 75 mg/m^2 every three week (q3w) until disease progression, unacceptable toxicity or death. Dose modifications were according to the locally approved label. Participants randomized to receive docetaxel had to be premedicated with corticosteroids according to local practice.
  Arms: Docetaxel
Drug: Atezolizumab — Participants received atezolizumab of 1200 mg (equivalent to an average body weight-based dose of 15 milligram per kilogram [mg/kg]) which was administered by IV infusion q3w on Day 1 of each 21 day cycle. Participants were allowed to continue treatment beyond progression per response evaluation criteria in solid tumors (RECIST) v1.1 if they were experiencing clinical benefit per investigator, did not have a decline in performance status, did not have signs or symptoms of unequivocal progression, did not have tumor progression at critical sites, and signed an informed consent signature page acknowledging deferment any standard treatment options that may exist in favor of continuing atezolizumab.
  Arms: Atezolizumab

SUMMARY:
This multicenter, open-label, randomized study will evaluate the efficacy and safety of Atezolizumab compared with docetaxel in participants with advanced or metastatic non-small cell lung cancer after platinum failure. Participants will be randomized to receive either Atezolizumab 1200 milligram (mg) intravenously every 3 weeks or docetaxel 75 milligram per meter square (mg/m^2) intravenously every 3 weeks. Treatment with Atezolizumab may be continued as long as participants are experiencing clinical benefit as assessed by the investigator, i.e., in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Locally advanced or metastatic (Stage IIIB, Stage IV, or recurrent) non-small cell lung cancer (NSCLC)
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens
* Disease progression during or following treatment with a prior platinum-containing regimen for locally advanced, unresectable/inoperable or metastatic NSCLC or disease recurrence within 6 months of treatment with a platinum-based adjuvant/neoadjuvant regimen
* Measurable disease, as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Known active or untreated central nervous system (CNS) metastases as determined by CT or MRI evaluation during screening and prior radiographic assessments
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active hepatitis B or hepatitis C
* Prior treatment with docetaxel
* Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (65):
- United States (29):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente - San Marcos, San Marcos, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Centers - Colorado Springs (Circle), Lone Tree, Colorado
  - Ocala Oncology Center, Ocala, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - New England Cancer Specialists, Scarborough, Maine
  - Karmanos Cancer Institute.., Detroit, Michigan
  - Billings Clinic; Research Center, Billings, Montana
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - The Valley Hospital, Paramus, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Broome Oncology - Binghamton, Binghamton, New York
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Center for Biomedical Research LLC, Knoxville, Tennessee
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- Belgium (2):
  - UZ Leuven Gasthuisberg, Leuven
  - Chr de La Citadelle, Liège
- Canada (2):
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- France (5):
  - Hopital Gabriel Montpied; Service de Pneumologie, Clermont-Ferrand
  - Hôpital Nord Michallon; Pneumologie, La Tronche
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Centre Hospitalier de Saint Brieuc - Hôpital Yves Le Foll; Pneumologie, Saint-Brieuc
  - Hopital Larrey; Pneumologie, Toulouse
- Germany (4):
  - Asklepios-Fachkliniken Muenchen-Gauting; Onkologie, Gauting
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin II, Halle
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Universitätsklinikum Regensburg; Klinik und Poliklinik für Innere Medizin II, Pneumologie, Regensburg
- Italy (2):
  - Citta Ospedaliera; Divisione Oncologia Medica, Avellino, Campania
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Woj.Wielospecjalistyczne Centrum Onkologii i Traumatologii; Oddz.Hematologii Pododz.Chemioterapii, Lodz
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy; Oddzial Iii, Otwock
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- South Korea (3):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
- Spain (4):
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Universitetssjukhuset Linköping; Lungmedicinkliniken, Linköping, Sweden
- Thailand (3):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Rajavithi Hospital; Division of Medical Oncology, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
- Turkey (Türkiye) (2):
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
- United Kingdom (4):
  - Royal Free Hospital; Dept of Oncology, London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Charing Cross Hospital; Medical Oncology., London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester

REFERENCES:
- [Derived] Dong Y, Zhu Y, Zhuo M, Chen X, Xie Y, Duan J, Bai H, Hao S, Yu Z, Yi Y, Guan Y, Yuan J, Xia X, Yi X, Wang J, Wang Z. Maximum Somatic Allele Frequency-Adjusted Blood-Based Tumor Mutational Burden Predicts the Efficacy of Immune Checkpoint Inhibitors in Advanced Non-Small Cell Lung Cancer. Cancers (Basel). 2022 Nov 17;14(22):5649. doi: 10.3390/cancers14225649. PMID 36428744
- [Derived] Shemesh CS, Chan P, Legrand FA, Shames DS, Das Thakur M, Shi J, Bailey L, Vadhavkar S, He X, Zhang W, Bruno R. Pan-cancer population pharmacokinetics and exposure-safety and -efficacy analyses of atezolizumab in patients with high tumor mutational burden. Pharmacol Res Perspect. 2020 Dec;8(6):e00685. doi: 10.1002/prp2.685. PMID 33241650
- [Derived] Chalabi M, Cardona A, Nagarkar DR, Dhawahir Scala A, Gandara DR, Rittmeyer A, Albert ML, Powles T, Kok M, Herrera FG; imCORE working group of early career investigators. Efficacy of chemotherapy and atezolizumab in patients with non-small-cell lung cancer receiving antibiotics and proton pump inhibitors: pooled post hoc analyses of the OAK and POPLAR trials. Ann Oncol. 2020 Apr;31(4):525-531. doi: 10.1016/j.annonc.2020.01.006. Epub 2020 Jan 16. PMID 32115349
- [Derived] Fehlings M, Jhunjhunwala S, Kowanetz M, O'Gorman WE, Hegde PS, Sumatoh H, Lee BH, Nardin A, Becht E, Flynn S, Ballinger M, Newell EW, Yadav M. Late-differentiated effector neoantigen-specific CD8+ T cells are enriched in peripheral blood of non-small cell lung carcinoma patients responding to atezolizumab treatment. J Immunother Cancer. 2019 Sep 12;7(1):249. doi: 10.1186/s40425-019-0695-9. PMID 31511069
- [Derived] Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, Park K, Smith D, Artal-Cortes A, Lewanski C, Braiteh F, Waterkamp D, He P, Zou W, Chen DS, Yi J, Sandler A, Rittmeyer A; POPLAR Study Group. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1837-46. doi: 10.1016/S0140-6736(16)00587-0. Epub 2016 Mar 10. PMID 26970723

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 527 participants were screened, of whom 287 participants were randomized. 143 participants to the docetaxel arm and 144 participants to the atezolizumab arm. Overall, 10 participants (8 in the docetaxel arm and 2 in the atezolizumab arm) did not receive any study treatment.
Groups:
- Docetaxel: Participants received docetaxel 75 milligram per squared meters (mg/m^2) administered intravenously on Day 1 of each 21 day cycle until disease progression or unacceptable toxicity or death.
Period: Overall Study
Arm/Group | Docetaxel | Atezolizumab
Started | 143 | 144
Received Treatment (Two patients in the docetaxel arm crossed over to receive atezolizumab treatment.) | 135 | 142
Completed (Study terminated by Sponsor participants either discontinued or enrolled in extension study) | 0 | 0
Not Completed | 143 | 144
Not completed — Death | 118 | 121
Not completed — Withdrawal by Subject | 15 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Study Terminated by Sponsor | 8 | 14
Not completed — Terminated by Sponsor After 31 Aug 2018 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population for efficacy analyses included all randomized participants, regardless of whether they received any study drug. In the efficacy analyses, the ITT population, participants were grouped according to the treatment arm to which they were assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel | Atezolizumab | Total
Number analyzed (Participants) | 143 | 144 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.4) | 61.5 (9.2) | 61.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 51 | 118
  Male | 76 | 93 | 169

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause. Data for participants who were not reported as dead at the time of analysis was censored at the date when they were last known to be alive.
Time Frame: From the time of randomization to the date of death due to any cause or up to data cut off date: 01 Dec 2015 (up to 28 months)
Population: ITT population for efficacy analyses included all randomized participants, regardless of whether they received any study drug. In the efficacy analyses, the ITT population, participants were grouped according to the treatment arm to which they were assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 143 | 144
months | 9.7 [8.6 to 12.0] | 12.6 [9.7 to 16.0]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; Hazard ratios (HR) were estimated by a Cox regression model; Test type: Superiority or Other; p = 0.0106, Log rank (Stratified); Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.52 to 0.92]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with confirmed objective tumor response, complete response (CR) or partial response (PR), as determined by investigator using RECIST v1.1 criteria. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Baseline until date of death due to any cause or up to data cut off date: 01 Dec 2015 (up to 28 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 143 | 144
percentage of participants | 14.7 [9.33 to 21.57] | 15.3 [9.83 to 22.21]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; Test type: Superiority or Other; p = 0.8884, Cochran-Mantel-Haenszel; Difference in Response Rates = 0.59, 95% CI 2-sided [-7.67 to 8.85]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time (in months) between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using response evaluation criteria In solid tumors (RECIST) v1.1. Progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions including baseline In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 143 | 144
months | 3.4 [2.8 to 4.1] | 2.7 [2.0 to 4.1]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; HR were estimated by a Cox regression model. The two treatment comparison was based on a stratified log-rank test; Test type: Superiority or Other; p = 0.5563, Log rank (Stratified); Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.71 to 1.20]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the duration from the first tumor assessment that supports the participant's objective response (CR or PR, whichever is first recorded) to disease progression or death due to any cause, whichever occurs first.
Time Frame: as for outcome 1
Population: ITT population for efficacy analyses included all randomized participants, regardless of whether they received any study drug. Here, number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 21 | 21
months | 7.2 [5.6 to 12.5] | 18.6 [11.6 to NA] — Upper limit of confidence interval (CI) was not achieved due to low number of participants with event.
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; HR were estimated by a unstratified Cox regression model; Test type: Superiority or Other; p = 0.0028, Log rank (unstratified); Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.15 to 0.70]

5. Secondary Outcome: ORR (Modified RECIST)
Description: ORR was defined as the percentage of participants with confirmed objective tumor response, CR or PR, as determined by investigator using modified RECIST criteria. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to l< 10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From the time of randomization to the date of death due to any cause or up to data cut off date: 08 May 2015 (up to 21 months)
Population: ITT population for efficacy analyses included all randomized participants, regardless of whether they received any study drug. In the efficacy analyses, the ITT population, participants were grouped according to the treatment arm to which they were assigned. The data was planned to be reported for Atezolizumab arm only
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 144
percentage of participants | 16.7 [10.98 to 23.78]

6. Secondary Outcome: PFS (Modified RECIST)
Description: PFS was defined as the time (in months) between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using modified RECIST criteria. PD: at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 144
months | 4.2 [3.9 to 6.9]

7. Secondary Outcome: DOR (Modified RECIST)
Description: as for outcome 4
Time Frame: as for outcome 5
Population: ITT population for efficacy analyses included all randomized participants, regardless of whether they received any study drug. Here, number of participants analyzed signifies the number of participants who were evaluable for this outcome measure. The data was planned to be reported for Atezolizumab arm only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 24
months | 14.9 [11.6 to NA] — Upper limit of CI was not achieved due to low number of participants with event.

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 31 August 2018
Description: Treatment-emergent adverse events are reported here and they include all adverse events that occurred on or after first dose of study drug until 30 days after last administration of study drug or initiation of another non-protocol anti-cancer therapy after the last administration of study drug, or clinical data cutoff date, whichever occurs first. Adverse Events reporting is for the Safety Evaluable Population, defined as patients who received any amount of any component of study treatment.
Arm/Group | Docetaxel | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 118/143 | 121/144
Serious Adverse Events (participants affected / at risk) | 46/135 | 53/142
Other Adverse Events (participants affected / at risk) | 125/135 | 127/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=135) | Atezolizumab (N=142)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (2) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 10 (13)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (5) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Contrast Media Allergy (Immune system disorders) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Thoracic Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Device Dislocation (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=135) | Atezolizumab (N=142)
Hypotension (Vascular disorders) | 4 (4) | 9 (9)
Asthenia (General disorders) | 22 (28) | 16 (26)
Chest pain (General disorders) | 6 (8) | 12 (13)
Fatigue (General disorders) | 55 (87) | 55 (82)
Oedema peripheral (General disorders) | 13 (18) | 9 (11)
Pain (General disorders) | 10 (11) | 6 (7)
Pyrexia (General disorders) | 16 (19) | 23 (28)
Insomnia (Psychiatric disorders) | 11 (12) | 24 (26)
Weight decreased (Investigations) | 11 (11) | 20 (24)
Anaemia (Blood and lymphatic system disorders) | 27 (38) | 28 (53)
Neutropenia (Blood and lymphatic system disorders) | 15 (23) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (40) | 45 (61)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (32) | 35 (41)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 11 (12)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 15 (21)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (14)
Dizziness (Nervous system disorders) | 11 (12) | 10 (16)
Headache (Nervous system disorders) | 10 (10) | 15 (18)
Neuropathy peripheral (Nervous system disorders) | 17 (21) | 4 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (21) | 1 (2)
Lacrimation increased (Eye disorders) | 7 (9) | 1 (1)
Constipation (Gastrointestinal disorders) | 32 (34) | 32 (33)
Diarrhoea (Gastrointestinal disorders) | 38 (51) | 25 (38)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 8 (12)
Nausea (Gastrointestinal disorders) | 45 (64) | 32 (45)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 3 (3)
Vomiting (Gastrointestinal disorders) | 18 (20) | 20 (26)
Alopecia (Skin and subcutaneous tissue disorders) | 52 (57) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (6)
Nail disorder (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 16 (26)
Rash (Skin and subcutaneous tissue disorders) | 16 (19) | 15 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 23 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 21 (22)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 9 (13)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 20 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (24) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (19) | 10 (12)
Hypothyroidism (Endocrine disorders) | 0 (0) | 13 (14)
Decreased appetite (Metabolism and nutrition disorders) | 29 (37) | 51 (60)
Dehydration (Metabolism and nutrition disorders) | 11 (11) | 6 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 9 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 9 (15)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 12 (17)
Influenza like illness (General disorders) | 2 (2) | 8 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (7) | 10 (15)
Chills (General disorders) | 4 (4) | 8 (9)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 8 (16)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 10 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.